CLINICAL TRIAL: NCT06606145
Title: Influence of the Microsugical Treatment (by Free Node Transfer And/or Lympho-venous Anastomosis (LVA)) of Secondary Lymphedema Following Axillary Lymph Node Dissection or Sentinel Node Biopsy, on the Health Related Quality of Life, Limb Volume Change, Subcutal and Dermal Thickness
Brief Title: Reduction of Arm Volume and Improvement in Lymphedema Via Surgery
Acronym: REFRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Moustapha Hamdi, Prof. Dr. Moustapha Hamdi, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUN 143201316894
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Lymphedema; Lymphedema Arm; Lymphedema of Arm; Lymphedema of Upper Limb; Lymphedema, Secondary
Keywords: lymphedema; lymphovenous anastomosis; vascularized lymph node transplant; LVA; VLNT
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lymphovenous Anastomoses (LVA) (Experimental): Patients with BCRL recieve one ore more Lymphovenous Anastomoses (LVA) on the affected limb. This involves connecting functional lymphatic vessels to nearby veins, allowing for the rerouting of lymphatic fluid into the venous system, thus improving lymphatic drainage. All patients had CDT pre- and post-op.
  Interventions: Procedure: Lymphovenous Anastomosis
- Vascularized Lymph Node Transfer (VLNT) (Experimental): Patients with BCRL recieve a Vascularized Lymph Node Transfer (VLNT) on the affected limb. This involves transferring healthy lymph nodes along with their blood supply to the affected lymphoedematous area, aiding in lymphatic fluid transport and potentially promoting lymphangiogenesis. All patients had CDT pre- and post-op.
  Interventions: Procedure: Vascularized Lymph Node Transfer
- LVA + VLNT (Experimental): Patients with BCRL recieve a combined simultaneous surgical intervention during which both VLNT and one or more LVA are performed on the affected limb. All patients had CDT pre- and post-op.
  Interventions: Procedure: Combined Lymphovenous Anastomosis and Vascularized Lymph Node Transfer
- Complex Decongestive Therapy (CDT) (Active Comparator): Patients with BCRL who refuse to undergo further surgical treatment after breast cancer surgery are offered conservative therapy. The current standard of care for most BRCL patients includes conservative measures known as Complex Decongestive Therapy (CDT) consisting of compression therapy with low-stretch bandages, manual lymphatic drainage, exercise, and skincare.
  Interventions: Procedure: Complex Decongestive Therapy

INTERVENTIONS:
Procedure: Lymphovenous Anastomosis — LVA involves connecting functional lymphatic vessels to nearby veins, allowing for the rerouting of lymphatic fluid into the venous system, thus improving lymphatic drainage.
  Other Names: LVA; Lymphovenous Bypass; LVB; Lymphaticovenous Anastomosis; Lymphatico-venous Anastomosis
  Arms: Lymphovenous Anastomoses (LVA)
Procedure: Vascularized Lymph Node Transfer — VLNT involves transferring healthy lymph nodes along with their blood supply to the affected lymphoedematous area, aiding in lymphatic fluid transport and potentially promoting lymphangiogenesis.
  Other Names: VLNT; Lymph Node Transfer; Lymph Node Transplant; Vascularized Lymph Node Transplant
  Arms: Vascularized Lymph Node Transfer (VLNT)
Procedure: Combined Lymphovenous Anastomosis and Vascularized Lymph Node Transfer — Combined simultaneous surgical intervention during which both VLNT and LVA are performed on the operated limb.
  Other Names: LVA + VLNT; LVA & VLNT
  Arms: LVA + VLNT
Procedure: Complex Decongestive Therapy — The current standard of care for most BRCL patients includes conservative measures known as Complex Decongestive Therapy (CDT), consisting of compression therapy with low-stretch bandages, manual lymphatic drainage, exercise, and skincare.
  Other Names: CDT
  Arms: Complex Decongestive Therapy (CDT)

SUMMARY:
This clinical trial aims to evaluate the effectiveness of lymphatic microsurgical treatments in reducing limb volume in female patients with breast cancer-related lymphedema (BCRL).

The study focuses on three treatments: Lymphovenous Anastomosis (LVA), Vascularized Lymph Node Transfer (VLNT), and Complex Decongestive Therapy (CDT).

The main questions it aims to answer are:

* Can LVA, VLNT, or their combination significantly reduce limb volume in patients with BCRL?
* How does the effectiveness of these surgical interventions compare to CDT alone?

Researchers will compare patients who undergo LVA, VLNT, or a combination of both to those receiving only CDT to determine the effectiveness of surgical interventions in reducing lymphedema symptoms.

Participants will:

* Undergo pre- and post-operative limb volume measurements.
* Receive either LVA, VLNT, or combined LVA and VLNT surgery, or continue CDT alone.
* Be monitored for one year to assess changes in limb volume and quality of life.

DETAILED DESCRIPTION:
This clinical trial aims to explore the effectiveness of surgical interventions for breast cancer-related lymphedema (BCRL), a chronic and often debilitating condition caused by lymphatic system damage following breast cancer treatments, such as lymph node dissection or radiation therapy. BCRL affects a significant proportion of breast cancer survivors, leading to arm swelling, discomfort, restricted mobility, and recurrent infections.

Standard management of BCRL includes conservative measures known as Complex Decongestive Therapy (CDT), which involves manual lymphatic drainage, compression therapy, exercise, and skincare. While CDT offers symptomatic relief, it does not address the underlying lymphatic dysfunction. In contrast, microsurgical procedures like Lymphovenous Anastomosis (LVA) and Vascularized Lymph Node Transfer (VLNT) are emerging as more definitive treatments for BCRL, targeting the lymphatic system itself.

LVA involves connecting small functional lymphatic vessels to nearby veins, allowing lymphatic fluid to bypass damaged lymph nodes and enter the venous system, improving drainage. It is particularly suited for patients with early-stage lymphedema (ISL stage I) where functional lymphatic vessels are still present.

VLNT involves transferring healthy lymph nodes along with their blood supply from a donor site (such as the groin or lateral thorax) to the affected area, promoting lymphangiogenesis and improving lymphatic transport. VLNT is more suitable for advanced stages of lymphedema (ISL stage II), where lymphatic vessels are more severely damaged.

The study will evaluate the outcomes of patients who undergo LVA, VLNT, or a combination of both, in comparison to a control group receiving only CDT. The surgical selection is based on preoperative imaging with indocyanine green (ICG) lymphography to assess the status of the lymphatic system. Each patient's lymphedema stage, severity, and individual characteristics are taken into consideration when choosing the most appropriate treatment.

Patients will be followed for one year postoperatively to measure the effectiveness of each treatment, with the primary outcome being limb volume reduction. Limb volume will be assessed using a perometer, an objective and reliable tool for measuring arm volume. Secondary outcomes include improvement in quality of life, frequency of infections, and the need for ongoing CDT post-surgery.

This study seeks to provide valuable insights into the comparative effectiveness of LVA, VLNT, and CDT in managing BCRL. While the benefits of microsurgical interventions are promising, particularly in reducing limb volume and infections, this trial aims to provide robust evidence to guide clinical decision-making and improve patient outcomes. By comparing different approaches, the study will help to clarify which surgical interventions are most beneficial for different stages of BCRL and establish clearer selection criteria for these treatments.

ELIGIBILITY:
Inclusion Criteria:

* at least one of the following persistent complaints of one of the upper extremities: heaviness, pain, recurrent infections

Exclusion Criteria:

* negative volume difference between affected and normal limb, bilateral mastectomy, bilateral axillary lymph node dissection (ALND), ongoing radio- and chemotherapy, ISL stage III, and receiving other simultaneous debulking procedures during lymphedema surgery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with Breast Cancer-Related Lymphedema (BCRL)
Enrollment: 179 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Relative interlimb difference | Before intervention and one year post-intervention
  Change in relative interlimb difference (RID) between the affected and contralateral limb

SECONDARY OUTCOMES:
Number of infection episodes after surgery | One year post-intervention
  The number of post-interventional erysipelas episodes is recorded for 12 months after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussel Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Anonymized individual participant data can be provided upon request by ICMJE journal editors.

REFERENCES:
- [Derived] Zeltzer AA, Nistor A, Adriaenssens N, Deleuze J, Giunta G, Hamdi M. Outcomes of Lymphovenous Anastomoses and Vascularized Lymph Node Transplant in the Combined Surgical Treatment of Lymphedema: A Prospective Cohort Study. Plast Reconstr Surg. 2026 Jan 1;157(1):163-175. doi: 10.1097/PRS.0000000000012326. Epub 2025 Jul 22. PMID 40707214